CLINICAL TRIAL: NCT07039318
Title: Mesenchymal Stem Cell Therapy in Diabetic Kidney Disease-A Double-blind, Placebo-controlled, Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Collaborators: Pak Emirates Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSC-CKD/2022
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Kidney Disease
Keywords: diabetic kidney disease; mesenchymal stem cells; randomized controlled trial
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is an interventional, double blind, randomized, controlled clinical trial where participants either receive mesenchymal stem cells (30 million cells) or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Mesenchymal stem cells (30 million cells)
  Interventions: Biological: Mesenchymal stem cells
- Normal Saline (Placebo) (Placebo Comparator): Normal Saline (Placebo)
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells
  Arms: Mesenchymal stem cells
Drug: Normal Saline (Placebo) — Normal Saline (Placebo)
  Arms: Normal Saline (Placebo)

SUMMARY:
Diabetes had global prevalence of 9% in 2014 and is increasing alarmingly, affecting approximately 387 million people worldwide. It is strongly linked to complications, like chronic kidney failure, blindness and neurdegeneration. From 1999-2006, prevalence of chronic kidney disease (CKD) stage 1-2 was 11.5%, and stage 3-4 was 58%, while its prevalence in Pakistan is 12.5%. CKD is a pathophysiological process with multiple etiologies, eventually resulting in irreversible nephron damage and leading to End Stage Renal Disease (ESRD), rendering the patient permanently dependent on Renal Replacement. In Pakistan, the prevalence of diabetic ESRD is 22%. Only supportive management is offered, resulting in either dialysis dependency or transplant. High CKD prevalence, renal replacement therapy and associated morbidity-mortality demands more effective and easier treatment option. We propose Mesenchymal Stem Cells (MSC) therapy for reversing the chronic kidney damage caused by type2 diabetes.

DETAILED DESCRIPTION:
Diabetes cases increased from 108 million in 1980 to 422 million in 2014 worldwide. Its prevalence has risen more rapidly in low- and middle-income countries than in high-income countries. It has become the leading cause of blindness, kidney failure, heart attacks, stroke and amputation of lower limbs. Damage to kidneys due to high blood is a serious threat, over time they stop the filtration process blood, leading to Chronic Kidney Disease. Approximately 1 in 3 adults with diabetes has CKD, which leads to kidney failure in worst cases and the only options left for the patient are regular dialysis or kidney transplant. Both these options are usually scarce, unaffordable and unavailable in developing countries like Pakistan. In finding an easier and effective treatment option for CKD secondary to diabetes it was found that MSCs can stop tissue damage progression in CKD, this has been extensively investigated in preclinical studies till now. Bone marrow derived MSCs are multipotent, including hematopoietic stem cell, mesenchymal stromal cells and endothelial progenitor cell. MSCs have anti-inflammatory and antifibrotic properties and can suppress maturation, activation and proliferation of T, B and NK cells in vitro and down regulate immune response in vivo. Beneficial effects of MSCs are seen largely through immunomodulatory and paracrine mechanisms like production of growth factors and cytokines with immunosuppressive, anti-inflammatory, anti-apoptotic and proliferative effects. Cultured MSCs release large amounts of pro-angiogenic factor; vascular endothelial growth factor which facilitates glomerular and tubular recovery. MSC therapy in CKD-preclinical studies have shown that single dose of bone marrow-derived MSCs in rats decreased interstitial fibrosis, tubular atrophy, T-cell and macrophage infiltration, and the expression of inflammatory cytokines. This has been attributed to their paracrine immunomodulatory properties rather than long-term engraftment. MSCs also have the capacity to induce proliferation of renal glomerular and tubular cells and increase cellular survival. In preclinical studies injected MSCs secrete pro-angiogenic and trophic factors which enhance proliferation and decrease apoptosis of tubular cells. However, engraftment and trans-differentiation was not observed in the majority of the studies. Although there is a large gap between scientific knowledge and clinical translation for a safe and effective stem cell-based therapy, stem cells hold great promise for the treatment of CKD. We aim to study the efficacy of MSCs treatment in diabetic nephropathy CKD stage 2 and 3 due to type 2 Diabetes Mellitus. For this purpose, we have designed a randomized, double-blinded, placebo-controlled clinical trial to determine the efficacy of MSC therapy in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients between 18 and 75 years of age having Type-2 Diabetes with CKD stage 2,3 and 4: (eGFR 15-90 mL/min/1.73 m2).

Exclusion Criteria:

Patients with a history of other comorbidities like previous myocardial infarction, pulmonary disease, pregnant females, unable to follow or return for evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
isotopic DTPA Scan | To be carried out at enrollment and at six months' post-intervention
  Glomerular Filtration Rate using Renal isotope 99mTc-DTPA

SECONDARY OUTCOMES:
Glycosylated Hemoglobin level | To be carried out at baseline and at six months post-intervention
  Glycosylated Hemoglobin using HBA1c level in blood

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - National Institute of Blood and Marrow Transplant (NIBMT), Pakistan/Armed Forces Bone Marrow Transplant Centre, Rawalpindi
  - Pak Emirates Military Hospital, Rawalpindi (PEMH), Rawalpindi

IPD SHARING:
Plan to Share IPD: Undecided